CLINICAL TRIAL: NCT01828060
Title: Efficacy of Jobelyn™ Consumption on Hemoglobin Levels in a Borderline Anemic Population.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Principal Investigator, Gitte Jensen, Ph.D., Research director, Natural Immune Systems Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NIS8914; NIS8914 (Other Grant/Funding Number: Health Forever Product Limited. Lagos, Nigeria)
Record Dates: First submitted 2013-04-02; First posted 2013-04-10 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Jobelyn™ (Experimental): Dietary supplement Jobelyn™, 500mg daily for 8 weeks Jobelyn is a sorghum bicolor extract marketed as dietary supplement Other Name: Sorghum bicolor extract
  Interventions: Dietary Supplement: Jobelyn™
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Jobelyn™ — Sorghum bicolor leaf sheath extract
  Arms: Jobelyn™
Dietary Supplement: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the timing and magnitude of improvements to red blood cell health associated with consumption of Jobelyn™.

DETAILED DESCRIPTION:
From past history, case studies in Nigeria, as well as testimonials from all over the world, have shown a robust increase in hemoglobin within a few weeks in people with serious cases of anemia present under disease conditions such as sickle cell, Malaria, HIV, or cancer. In parallel, improvements in red blood cell health were also seen in many healthy people with general low blood counts due to undetermined factors.

A clinical study on anemia is currently ongoing in Nigeria. The study population is focused on women and aims at evaluating whether Jobelyn™ consumption can help increase hemoglobin and thus reduce risk factors associated with gynecological surgery in a Nigerian cohort of gynecological patients (ClinicalTrials.gov Identifier: NCT01670955).

As a parallel to the ongoing study in Nigeria, this study protocol will help to systematically examine the effects of Jobelyn™ on anemic conditions in an otherwise healthy North American population, and help document the speed and magnitude of improvements in a population without concomitant infections or sickle cell anemia.

Twenty-four human subjects of both genders will be tested over a period of 8 weeks. Both genders may enroll in the study, but we expect more women to be eligible, due to effects of menses and prolonged consumption of birth control pills. Recruiting of volunteers will happen via NIS Labs. A screening blood draw will be used for CBC/differential and the hemoglobin level help determine eligibility.

Enrolled subjects will randomized to consume placebo or Jobelyn™ for 8 weeks, during which time subjects are monitored at baseline, and after 3 days, 7 days, and 2, 4, and 8 weeks. A fasting blood sample will be taken at each visit, and used for hemoglobin and fasting glucose measurements.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 year old people of either gender
* Borderline anemic (This is compensated for altitude of study location):
* Hemoglobin level at or below 13.5 g/dL(women)
* Hemoglobin level at or below 15.5 g/dL(men)

Exclusion Criteria:

* Known diagnosis with pernicious or other megaloblastic anemias, aplastic, sickle cell, thalassemia, autoimmune hemolytic anemias;
* Known diagnosis with Hashimoto's Disease;
* Known chronic kidney disease;
* Rheumatoid arthritis;
* Splenectomy;
* Serious active illness within past 12 months;
* Active cancer and/or chemotherapy within the last 12 months;
* Major surgery during past 8 weeks;
* Scheduled surgery during study;
* Received blood transfusion during the past 8 weeks;
* Having donated blood for 6 weeks prior to study, or planning to donate blood during the 8 week study;
* Distance athlete;
* Unable to commit to staying on a constant regimen of medication and supplements for the duration of the study, with the exception of changes to medication needed for optimal care;
* Changes to prescription medication within 2 weeks before starting the study;
* Participation in other clinical trials during the month before this study begins;
* Participating in other clinical trials during this study;
* Current use of any dietary supplements that may affect hemoglobin levels; Vitamin B12 (over 500 mcg), Iron (over 100mg), or any other dietary supplement that, in the opinion of the investigator, may affect hemoglobin levels;
* Currently experiencing intense stressful events/ life changes that would negatively affect compliance;
* Previous major gastrointestinal surgery (absorption of test product may be altered) (minor surgery is not a problem, including appendix and gallbladder removal);
* Females of child-bearing potential: Pregnant, nursing, or trying to become pregnant;
* Food allergies related to sorghum or rice.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Hemoglobin | 8 weeks
  Change in hemoglobin levels

SECONDARY OUTCOMES:
Fasting blood glucose | 8 weeks
  Change in fasting glucose levels

CONTACTS AND LOCATIONS:
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States

REFERENCES:
- [Background] Geera B, Ojwang LO, Awika JM. New highly stable dimeric 3-deoxyanthocyanidin pigments from sorghum bicolor leaf sheath. J Food Sci. 2012 May;77(5):C566-72. doi: 10.1111/j.1750-3841.2012.02668.x. Epub 2012 Apr 10. PMID 22489620
- [Background] Kayode AP, Nout MJ, Linnemann AR, Hounhouigan JD, Berghofer E, Siebenhandl-Ehn S. Uncommonly high levels of 3-deoxyanthocyanidins and antioxidant capacity in the leaf sheaths of dye sorghum. J Agric Food Chem. 2011 Feb 23;59(4):1178-84. doi: 10.1021/jf103963t. Epub 2011 Jan 25. PMID 21322653
- [Background] Camargo Filho I, Cortez DA, Ueda-Nakamura T, Nakamura CV, Dias Filho BP. Antiviral activity and mode of action of a peptide isolated from Sorghum bicolor. Phytomedicine. 2008 Mar;15(3):202-8. doi: 10.1016/j.phymed.2007.07.059. Epub 2007 Sep 24. PMID 17890069
- [Background] Oladiji AT, Jacob TO, Yakubu MT. Anti-anaemic potentials of aqueous extract of Sorghum bicolor (L.) moench stem bark in rats. J Ethnopharmacol. 2007 May 22;111(3):651-6. doi: 10.1016/j.jep.2007.01.013. Epub 2007 Jan 18. PMID 17306481
- [Background] Falade OS, Otemuyiwa IO, Oladipo A, Oyedapo OO, Akinpelu BA, Adewusi SR. The chemical composition and membrane stability activity of some herbs used in local therapy for anemia. J Ethnopharmacol. 2005 Oct 31;102(1):15-22. doi: 10.1016/j.jep.2005.04.034. PMID 16039811
- [Background] Benson KF, Beaman JL, Ou B, Okubena A, Okubena O, Jensen GS. West African Sorghum bicolor leaf sheaths have anti-inflammatory and immune-modulating properties in vitro. J Med Food. 2013 Mar;16(3):230-8. doi: 10.1089/jmf.2012.0214. Epub 2013 Jan 5. PMID 23289787